CLINICAL TRIAL: NCT02374346
Title: Factors Associated With the Presence of Postoperative Headache in Elective Surgery Patients: a Prospective Single Center Cohort Study
Brief Title: Postoperative Headache in Elective Surgery Patients
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Assistant Proffesor, Attikon Hospital
Other Study IDs: 8/11/2004
Record Dates: First submitted 2015-02-24; First posted 2015-02-27 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Drug Withdrawal Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the association of anaesthesia and surgery with postoperative headache in elective surgery patients By multiple logistic regression analysis of data collected during a six-month period from 446 patients undergoing elective surgery, a prospective single centre cohort study in a university hospital. Participants were interviewed preoperatively and for five days postoperatively regarding the appearance of headache; while demographics, life style, type of anaesthesia and surgery, the anaesthetic drugs administered and intraoperative adverse effects in elective surgery patients are recorded.

DETAILED DESCRIPTION:
A dedicated team interviewed patients preoperatively and during the first five postoperative days and collected data regarding medical history, surgery, anaesthesia and the presence of postoperative headache by manual record review. The frequency of preoperative headache was assessed by asking the subjects on the appearance or not of headache within the last year. Additional information were obtained to distinguish migraine which was deemed present only when the participants reported two or more of the following specific symptoms supporting this diagnosis as proposed by the International Headache Society; episodic headache (4-72 hours) with the following features: moderate or severe throbbing pain, worsened by movement, associated with nausea/vomiting, photophobia or phonophobia, with or without visual aura.

Specifically, preoperative data included patients' demographics, marital status, life-style and habits, as caffeine consumption (>200 mg/day or >2 cups of coffee/day), alcohol (drink equivalent > 15ml absolute alcohol) and tobacco consumption, previous experience or/and family history of headache. Intraoperative data included the type of anaesthesia (general, regional anaesthesia or their combination); anaesthetic drugs used; type and duration of surgery; intraoperative patients' position; and intraoperative adverse events including hypotension (decrease >20% from baseline), hypertension (increase >20% from baseline), hypercarbia (PaCO2 >6 kPa) and hypoxia (SpO2 <90%). Noticeably, the choice of anaesthetic technique and postoperative management were determined by the engaged anaesthesiologist.

Postoperative headache was defined as a dichotomous variable (i.e. present or not present) by asking the participants twice daily for the first five days (or less if discharged earlier) after anaesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients admitted in our hospital for elective general, orthopaedic, gynaecologic, ENT(ear nose and throat) and vascular procedures

Exclusion Criteria:

* patient refusal
* age under 18 years
* cognitive dysfunction
* head trauma or neurological disorders
* difficulty with language comprehension or any other inability to communicate verbally with the interviewer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients admitted in our hospital for elective general, orthopaedic, gynaecologic, ENT(ear nose and throat) and vascular procedures
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Elective Surgery Patients: A total number of 494 patients full fit the inclusion criteria and 446 completed the study (90.3 %).The 48 patients (9.7%) who did not complete the study were those operated or discharged during weekend.
Period: Overall Study
Arm/Group | Elective Surgery Patients
Started | 494
Completed | 446
Not Completed | 48
Not completed — operated or discharged during weekend | 48

BASELINE CHARACTERISTICS:
Population: A total number of 446 adult patients admitted for elective surgery were included in the study.
  Exclusion criteria: patient refusal, age under 18 years, cognitive dysfunction, head trauma or neurological disorders, difficulty with language comprehension or any other inability to communicate verbally with the interviewer.
Groups:
- Elective Surgery Patients: All adult patients admitted in our hospital for elective general, orthopaedic, gynaecologic, ear-nose-throat (ENT) and vascular procedures.
Arm/Group | Elective Surgery Patients
Number analyzed (Participants) | 446
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 396
  >=65 years | 50
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 321
  Male | 125
Region of Enrollment [Number; unit: participants]
  Greece | 446

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Postoperative Headache in Elective Surgery Patients
Description: The observed overall frequency of postoperative headache was 28.3% (N= 126) in the total sample.
Time Frame: 6 months
Population: Frequency of postoperative headache in total sample (n=446)," "Post-op Headache, no History of Headache (n=229)," "Post-op Headache, History of Headache (n=217), where n= number of participants analyzed"
Measure: Number; unit: participants
Groups:
- Elective Surgery Patients (Total Sample): postoperative headache in elective surgery patients
Arm/Group | Elective Surgery Patients (Total Sample)
Number analyzed (Participants) | 446
participants
  postoperative headache in total sample | 126
  postop headache with no history of headache | 37
  postop headache with previous history | 89

2. Secondary Outcome: Factors Associated With Postoperative Headache
Description: Demographic, anaesthetic and surgical factors associated with postoperative headache
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Postoperative Headache in the Total Sample: Factors for developing postoperative headache in the total number of participants
- Postoperative Headache Patients Without Headache History: Factors for developing postoperative headache in patients without previous history of headache.
Arm/Group | Postoperative Headache in the Total Sample | Postoperative Headache Patients Without Headache History
Number analyzed (Participants) | 446 | 218
participants
  female gender | 103 | 32
  sevoflurane administration | 91 | 27
  intraoperative hypotension | 98 | 23
  smoking | 79 | 22
  caffeine consumption | 104 | 34
Statistical Analysis 1: Comparison: Postoperative Headache in the Total Sample; Sevoflurane administration in developing postoperative headache; Test type: Non-Inferiority or Equivalence — Associations between categorical variables were tested by χ2 test, while differences between categorical and continuous variables were tested by Student's t test. Univariate analysis was performed with the computation of unadjusted odds ratios with 95% confidence intervals. A stepwise multiple logistic regression analysis was conducted to find independent factors; p = 0.001, t-test, 2 sided; Odds Ratio (OR) = 3.23, 95% CI 2-sided [2.04 to 5.13]
Statistical Analysis 2: Comparison: Postoperative Headache in the Total Sample; Smoking as a factor for developing postoperative headache; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.006, t-test, 2 sided; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.19 to 2.84]
Statistical Analysis 3: Comparison: Postoperative Headache in the Total Sample; Intraoperative hypotension associated with postoperative headache in total sample; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.008, t-test, 2 sided; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.22 to 3.66]
Statistical Analysis 4: Comparison: Postoperative Headache in the Total Sample; Female gender as a factor for developing postoperative headache; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.024, t-test, 2 sided; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.08 to 3.15]
Statistical Analysis 5: Comparison: Postoperative Headache Patients Without Headache History; Association of female gender and postoperative headache; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.005, t-test, 2 sided; Odds Ratio (OR) = 4.56, 95% CI 2-sided [1.58 to 13.17]
Statistical Analysis 6: Comparison: Postoperative Headache Patients Without Headache History; Association of intraoperative hypotension and postoperative headache; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.006, t-test, 2 sided; Odds Ratio (OR) = 3.79, 95% CI 2-sided [1.48 to 9.72]
Statistical Analysis 7: Comparison: Postoperative Headache Patients Without Headache History; Association of caffeine consumption and postoperative headache; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.041, t-test, 2 sided; Odds Ratio (OR) = 3.86, 95% CI 2-sided [1.06 to 14.06]
Statistical Analysis 8: Comparison: Postoperative Headache Patients Without Headache History; Association of sevoflurane administration and postoperative headache; Test type: Non-Inferiority or Equivalence — Associations between categorical variables were tested by χ2 test, while differences between categorical and continuous variables were tested by Student's t test.Univariate analysis was performed with the computation of unadjusted odds ratios with 95% confidence intervals. A stepwise multiple logistic regression analysis was conducted to find independent factors; p = 0.001, t-test, 2 sided; Odds Ratio (OR) = 4.26, 95% CI 2-sided [1.82 to 9.95]

ADVERSE EVENTS:
Description: Serious and Other [non-serious] adverse events were not collected/assessed
Arm/Group | Elective Surgery Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No